CLINICAL TRIAL: NCT04212208
Title: Pain Assessment in the Perioperative Area During IV Cannulation Using a Combination of EMLA and Low-frequency USG Probe Versus a Combination of EMLA Cream and High-frequency Probe in Pediatric Cases- A Randomized Control Trial
Brief Title: Pain Assessment in the Perioperative Area
Acronym: EMLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences, Rishikesh (Other Government)
Responsible Party: Principal Investigator, ADABALA VIJAY BABU, PRINCIPLE INVESTIGATOR, All India Institute of Medical Sciences, Rishikesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Pain, Procedural
MeSH Terms: conditions — Pain, Procedural | interventions — Catheterization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): EMLA cream + High-frequency USG probe kept for 15minutes.After 15 minutes IV cannulation will be done and Pain intensity assessment will be done using Faces Pain Scale-Revised (FPS-R)
  Interventions: Device: IV cannulation
- Control group (Active Comparator): EMLA cream+Low frequency USG probe kept over the cream for 15 minutes. IV cannulation will be done and Pain intensity assessment will be done using Faces Pain Scale-Revised (FPS-R)
  Interventions: Device: IV cannulation

INTERVENTIONS:
Device: IV cannulation — IV cannulation in the preoperative period

SUMMARY:
This study is mainly focusing on reducing the pain scores during IV cannulation in pediatric population in the preoperative period. Applying EMLA cream is a well-known fact world wide. we would like to study the effect of ultrasound waves in the penetration of the given drung into the skin so that we could achieve the effect of the drug quickly.

DETAILED DESCRIPTION:
To assess the intensity of pain in children in the perioperative area during IV cannulation using a combination of EMLA cream and low-frequency USG probe. To assess the intensity of pain in children in the perioperative area during IV cannulation using a combination of EMLA cream and high-frequency USG probe and final comparison between these groups will assess the effect of ultrasound in the penetration of the drug into the skin.

ELIGIBILITY:
Inclusion Criteria:

* All children in the preoperative period.

Exclusion Criteria:

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-26 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare the intensity of pain among control versus interventional groups. Pain intensity assessment will be done using Faces Pain Scale-Revised (FPS-R) | 15minutes
  to check the efficacy of high-frequency ultrasound probe in comparison to low-frequency probe in aiding the drug penetration there by decreasing the pain intensity during IV cannulation

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Adabala, MD, Study Chair — AIIMS Rishikesh
Locations (1):
- AIIMS, Rishikesh, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lucas VS, Burk RS, Creehan S, Grap MJ. Utility of high-frequency ultrasound: moving beyond the surface to detect changes in skin integrity. Plast Surg Nurs. 2014 Jan-Mar;34(1):34-8. doi: 10.1097/PSN.0000000000000031. PMID 24583666